CLINICAL TRIAL: NCT01479218
Title: Safety and Effectiveness Study With a New PDA Occluder for Closure of Patent Ductus Arteriosus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Occlutech International AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Occlutech-PDA1
Record Dates: First submitted 2011-11-18; First posted 2011-11-24 (Estimated); Last update posted 2024-02-15 (Actual); Status verified 2013-05

CONDITIONS: Patent Ductus Arteriosus
MeSH Terms: conditions — Ductus Arteriosus, Patent

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PDA Occluder (Other): single arm
  Interventions: Device: Occlutech PDA occluder

INTERVENTIONS:
Device: Occlutech PDA occluder — Four different sizes of Occluders will be evaluated based on pre-assessment of PDA size.

SUMMARY:
The objective of the study is to investigate the safety, efficacy and clinical utility of the Occlutech PDA device for closure of patent ductus arteriosus of all types.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a demonstrated patent ductus arteriosus
2. Female or male
3. Belonging to any ethnic group
4. Age between > 6 months and 70 years
5. Body weight > 6 kg < 120 kg

Exclusion Criteria:

1. Associated congenital cardiac anomalies,
2. Body weight < 6 Kilograms

General exclusion criteria

* presence of a known coagulation disorder
* thrombus at the position allocated for the implantation
* a vein thrombosis in the blood vessels chosen for the introducing system
* an active infection
* Nitinol intolerance (nickel or titanium)
* contrast medium intolerance
* patients who have a vascular system which is too small to admit the required sheath
* patients with pulmonary hypertension and pulmonary-vascular resistance of >8 Woods Units or a lung - / systemic resistance (PR/SR) of >0.4.

Ages: 6 Months to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2011-11; Primary Completion 2014-02 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Successful closure of patent ductus arterious without evidence of any complication assessed by echocardiongram, ECG and X-ray 30 and 90 days after implant. | 3 months

SECONDARY OUTCOMES:
Successful closure without evidence of residual shunt after 1 year confirmed by echocariodgram. Safety: freedom of major adverse events i.e periherial embolism or endocarditits. | 30, 90, 180 and 360 days after implant

CONTACTS AND LOCATIONS:
Overall Officials: Ziyad M Hijazi, Professor, Study Chair — Rush University medical center, Chicago, USA; Alwi Mazeni, Dr, Principal Investigator — IJN Heart Institute, Kuala Lumpur, Malaysia; Viet Minh Tri Nguyen, Dr, Principal Investigator — Pediatric hospital no 2, Hochiminh city, Vietnam
Locations (2):
- IJN National Heart Institute, Kuala Lumpur, Malaysia
- Pediatric Hospital no 2, Hochiminh City, Vietnam